CLINICAL TRIAL: NCT04683133
Title: Association Between 3D Quantitative Angiography Based FFR and Luminal Obstruction as Detected by Optical Coherence Tomography (OCT): the FAST OCT Study
Brief Title: The FAST OCT Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Abbott (Industry); Pie Medical Imaging (Unknown)
Responsible Party: Principal Investigator, Joost Daemen, Interventional Cardiologist, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: The FAST OCT study
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Tomography, Optical Coherence; Myocardial Revascularization; NSTEMI - Non-ST Segment Elevation MI; Unstable Angina; Coronary Arteriosclerosis; 3D-angio-based FFR
Keywords: OCT; 3D-angio-based FFR; Coronary Arteriosclerosis; NST-ACS
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, international, no-randomized, single-arm, investigator-initiated study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single arm (Other): Optical coherence tomography evaluation of coronary arteries with intermediate to severe stenosis.
  Interventions: Diagnostic Test: Optical coherence tomography assessment

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography assessment — Optical coherence tomography assessment of coronary arteries with intermediate to severe stenosis

SUMMARY:
This trial is designed to associate angiography-based fractional flow reserve (3D-angio-based FFR) values with optical coherence tomography findings in pre- and post-percutaneous coronary intervention in patients with non-ST segment elevation acute coronary syndromes.

DETAILED DESCRIPTION:
Prospective, multicenter, international, no-randomized, single-arm, investigator-initiated study, enrolling up to 200 patients with intermediate to severe coronary stenosis (30-90% diameter stenosis) in patients presenting with NST-ACS requiring coronary angiography assessment.

Patients will receive ad-hoc OCT evaluation of the target vessels and offline 3D-angio-based FFR evaluation.

The primary study parameter is the association between 3D-angio-based FFR values and OCT detected minimum luminal area pre- and post-PCI

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Presenting with NST-ACS
* At least one coronary vessel with intermediate to severe coronary stenosis (30% to 90% by visual estimation or online QCA)
* Target vessel with a reference vessel diameter (RVD) ≥2.5 and ≤ 5.0 mm as assessed by QCA or visual estimation
* The patient is willing to participate in the study
* Target vessel suitable for OCT imaging

Exclusion Criteria:

* Target vessel with a distal Thrombolysis In Myocardial Infarction (TIMI) flow <3
* Target lesion located within 5.0 mm of vessel origin
* Severe tortuosity
* Chronic total occlusion of the target vessel
* Target lesion is located in or supplied by an arterial or venous bypass graft.
* Impaired renal function (eGFR <30ml/min) *
* Pregnant or breastfeeding patients *
* Patient has a known allergy to contrast medium *
* Contraindication for the use of nitrates *
* Life expectancy <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The association between 3D-angio-based FFR and OCT detected minimum luminal area pre- and post-PCI | 0 days
  The association between 3D-angio-based FFR and OCT detected minimum luminal area pre- and post-PCI

SECONDARY OUTCOMES:
The association between 3D-angio-based FFR values and OCT detected causes of luminal obstruction pre-PCI | 0 days
  The association between 3D-angio-based FFR values and OCT detected causes of luminal obstruction pre-PCI
The association between 3D-angio-based FFR values and OCT detected causes of luminal obstruction post-PCI | 0 days
  The association between 3D-angio-based FFR values and OCT detected causes of luminal obstruction post-PCI
Accuracy of 3D-angio-based FFR to detect intraluminal obstructions pre-PCI | 0 days
  Accuracy of 3D-angio-based FFR to detect intraluminal obstructions pre-PCI
Accuracy of 3D-angio-based FFR to detect intraluminal obstructions post-PCI | 0 days
  Accuracy of 3D-angio-based FFR to detect intraluminal obstructions post-PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No